CLINICAL TRIAL: NCT01044407
Title: Developing a New, Dynamic, Therapeutic Pacemaker Algorithm for Stabilising Periodic Breathing in Chronic Heart Failure.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Darrel Francis, Imperial College
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: P10678
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2010-01-25 (Estimated); Status verified 2010-01

CONDITIONS: Periodic Breathing
Keywords: respiration; sleep apnea; pacemaker
MeSH Terms: conditions — Respiratory Aspiration; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pacemaker manipulation — Alternation of cardiac output by modulation of heart rate, atrioventricular delay and modulation from biventricular pacing to right ventricular pacing (where applicable)via a cardiac pacemaker

SUMMARY:
To evaluate whether cardiac output manipulation via a cardiac pacemaker can stabilise ventilation.

DETAILED DESCRIPTION:
Many patients with heart failure exhibit a distinctive abnormal cyclical breathing pattern, 'periodic breathing'. This means that patients have a worse prognosis and they have debilitating symptoms including breathlessness, fatigue and disrupted sleep. Many of these patients also have cardiac pacemakers fitted, to improve their heart function. We have discovered a new physiological mechanism linking the heart and lungs, and have shown that by changing the programmed settings of a cardiac pacemakers, we can change a patient's breathing. If we increase the programmed pacing heart rate, we increase the rate of delivery of carbon dioxide to the lungs temporarily, which increases ventilation. When we reduce the programmed pacing heart rate, the converse happens. We aim to demonstrate this phenomenon scientifically, and to use this information to stabilise periodic breathing in heart failure patients using pacemakers. We then plan to continue to investigate whether we can show that sleep quality is improved in heart failure patients with periodic breathing, by our pacing protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cardiac pacemakers implanted on standard clinical grounds, and either normal left ventricular systolic function (as assessed by echocardiogram) or impaired left ventricular systolic function and stable breathing patterns (as assessed by screening in outpatients' clinic).

Exclusion Criteria:

* Patients with atrial fibrillation with a ventricular rate of >70 bpm will be excluded.
* Patients with implantable cardiac defibrillators with anti-tachycardia therapy set at an unusually low rate (<120 bpm), because it would limit the ability to vary the heart rate during the experiment.
* Patients with significant respiratory disease (FEV1 <50% predicted) will be excluded, as will patients with any condition that who have any condition precluding them from lying comfortably on a bed for 90 minutes.
* Patients who have had a recent deterioration in condition i.e. admission in previous six weeks, those in a brittle condition and those who have end-stage renal failure requiring haemodialysis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-02 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
stability of ventilation | Per second

CONTACTS AND LOCATIONS:
Overall Officials: Darrel P Francis, MD, Principal Investigator — Imperial College London
Locations (1):
- Imperial NHS Trust, London, London, United Kingdom

REFERENCES:
- [Background] Baruah R, Manisty CH, Giannoni A, Willson K, Mebrate Y, Baksi AJ, Unsworth B, Hadjiloizou N, Sutton R, Mayet J, Francis DP. Novel use of cardiac pacemakers in heart failure to dynamically manipulate the respiratory system through algorithmic changes in cardiac output. Circ Heart Fail. 2009 May;2(3):166-74. doi: 10.1161/CIRCHEARTFAILURE.108.806588. Epub 2009 Mar 23. PMID 19808336